CLINICAL TRIAL: NCT02766829
Title: Comparison of Successful Spinal Needle Placement Between Crossed Leg Sitting Position and Traditional Sitting Position in Patients Underwent Urology Surgery
Brief Title: Comparison of Successful Spinal Needle Placement Between Crossed Leg Sitting Position and Traditional Sitting Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Sidharta K. Manggala, Consultant, Anesthesiologist, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes007
Record Dates: First submitted 2016-05-06; First posted 2016-05-10 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Adult Patients With Spinal Anesthesia
Keywords: spinal; anesthesia; sitting; cross leg; spinal-bone contact

ARMS (2):
- CLSP Group (Experimental): Those with cross leg sitting position: patients sit with both their knees flexed medially, hip flexed, resulting in pelvic leaning posteriorly and reducing lumbal lordosis.
  Interventions: Procedure: Cross leg sitting position
- TSP Group (Active Comparator): Those with traditional sitting position: patient is positioned with her knees flexed 90o, both feet hanging of the bed and propped up by a chair, both arms hugging a pillow, adducted pelvic, maximum pelvic flexion were done to create maximal sagittal lumbal flexion.
  Interventions: Procedure: Traditional sitting position

INTERVENTIONS:
Procedure: Cross leg sitting position — Subjects were set on cross leg sitting position before spinal anesthesia begun.
  Arms: CLSP Group
Procedure: Traditional sitting position — Subjects were set on traditional sitting position before spinal anesthesia begun.
  Arms: TSP Group

SUMMARY:
The study aimed to compare successful spinal needle placement between crossed leg sitting position and traditional sitting position in patients underwent urology surgery.

DETAILED DESCRIPTION:
Approval from Ethical Committee of Faculty of Medicine Universitas Indonesia was acquired prior conducting the study. Subjects were given informed consent before enrolling the study. Subjects were randomly divided into CLSP Group for crossed leg sitting position (n=105) and TSP Group for traditional sitting position (n=106). Non-invasive blood pressure (NIBP) monitor, eletrocardiography (ECG), oxygen nasal cannula and pulse-oxymetry was set on the subjects in the operation room. Baseline information was recorded. Spinal anesthesia was done by anesthesiology registrars that have done 50 spinal anesthesia procedures and have been explained about the protocol of spinal anesthesia injection in this study (to avoid bias). Outcome measures were the number of successful spinal needle placement in the first attempt, the difficulty level of landmark palpation for injection, and the number of needle-bone contact. Data was analyzed by SPSS (Statistical Package for Social Scientist) using Chi-Square test, Fisher Exact test, and Kolmogorov-Smirnov test. Significance value used was 5% with 80% power.

ELIGIBILITY:
Inclusion Criteria:

* subjects aged 18-60 years old-
* subjects with ASA physical status I-III who were planned to undergo urology surgery with spinal anesthesia
* Subjects who have been explained about the study, have agreed to enroll and have signed the informed consent form

Exclusion Criteria:

* uncooperative subjects
* subjects with relative and absolute contraindications to spinal anesthesia (coagulation disorders, thrombocytopenia, increases intracranial pressure, severe hypovolemia, severe heart valve disorders, local infection at the injection site, allergy toward local anesthetic agents, significant anatomical disorder of the spine, wound/scar on the lumbal area)
* subjects with body mass index (BMI) > 32 kg/m2

Drop out criteria:

* subjects who requestes to drop out of the study
* subjects in need of emergency treatment during spinal anesthesia procedure
* subjects with more than nine times redirected spinal needle (failed spinal anesthesia procedure).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 211 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
One shot successful spinal needle placement | 7 months
  The number of successful spinal needle placement in the first attempt
Needle-bone contact number | 7 months
  The number of needle-bone contact recorded.
The difficulty level of landmark palpation for injection | 7 months
  the difficulty level of landmark palpation for injection were assessed as easy or difficult.

SECONDARY OUTCOMES:
Spinal needle placement complications | 7 months
  Complications recorded were post dural puncture headache, low back pain and neural trauma.

CONTACTS AND LOCATIONS:
Overall Officials: Sidharta K Manggala, Consultant, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Central National Hospital, Jakarta, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Edwards ND, Callaghan LC, White T, Reilly CS. Perioperative myocardial ischaemia in patients undergoing transurethral surgery: a pilot study comparing general with spinal anaesthesia. Br J Anaesth. 1995 Apr;74(4):368-72. doi: 10.1093/bja/74.4.368. PMID 7734251
- [Background] Fettes PD, Jansson JR, Wildsmith JA. Failed spinal anaesthesia: mechanisms, management, and prevention. Br J Anaesth. 2009 Jun;102(6):739-48. doi: 10.1093/bja/aep096. Epub 2009 May 6. PMID 19420004
- [Background] Sprung J, Bourke DL, Grass J, Hammel J, Mascha E, Thomas P, Tubin I. Predicting the difficult neuraxial block: a prospective study. Anesth Analg. 1999 Aug;89(2):384-9. doi: 10.1097/00000539-199908000-00025. PMID 10439752
- [Background] Atallah MM, Demian AD, Shorrab AA. Development of a difficulty score for spinal anaesthesia. Br J Anaesth. 2004 Mar;92(3):354-60. doi: 10.1093/bja/aeh073. Epub 2004 Jan 22. PMID 14742333
- [Background] Kim JH, Song SY, Kim BJ. Predicting the difficulty in performing a neuraxial blockade. Korean J Anesthesiol. 2011 Nov;61(5):377-81. doi: 10.4097/kjae.2011.61.5.377. Epub 2011 Nov 23. PMID 22148085
- [Background] de Filho GR, Gomes HP, da Fonseca MH, Hoffman JC, Pederneiras SG, Garcia JH. Predictors of successful neuraxial block: a prospective study. Eur J Anaesthesiol. 2002 Jun;19(6):447-51. doi: 10.1017/s0265021502000716. PMID 12094920
- [Background] Chin KJ, Karmakar MK, Peng P. Ultrasonography of the adult thoracic and lumbar spine for central neuraxial blockade. Anesthesiology. 2011 Jun;114(6):1459-85. doi: 10.1097/ALN.0b013e318210f9f8. PMID 21422997
- [Background] Fisher KS, Arnholt AT, Douglas ME, Vandiver SL, Nguyen DH. A randomized trial of the traditional sitting position versus the hamstring stretch position for labor epidural needle placement. Anesth Analg. 2009 Aug;109(2):532-4. doi: 10.1213/ane.0b013e3181ac6c79. PMID 19608828
- [Background] Soltani Mohammadi S, Hassani M, Marashi SM. Comparing the squatting position and traditional sitting position for ease of spinal needle placement: a randomized clinical trial. Anesth Pain Med. 2014 Apr 5;4(2):e13969. doi: 10.5812/aapm.13969. eCollection 2014 May. PMID 24790901
- [Background] Watanabe S, Kobara K, Ishida H, Eguchi A. Influence of trunk muscle co-contraction on spinal curvature during sitting cross-legged. Electromyogr Clin Neurophysiol. 2010 Apr-Jun;50(3-4):187-92. PMID 20552952
- [Background] Biswas BK, Agarwal B, Bhattarai B, Dey S, Bhattacharyya P. Straight versus flex back: Does it matter in spinal anaesthesia? Indian J Anaesth. 2012 May;56(3):259-64. doi: 10.4103/0019-5049.98772. PMID 22923825
- [Background] Shankar H, Rajput K, Murugiah K. Correlation between spinous process dimensions and ease of spinal anaesthesia. Indian J Anaesth. 2012 May;56(3):250-4. doi: 10.4103/0019-5049.98769. PMID 22923823
- [Background] Purepong N, Jitvimonrat A, Boonyong S, Thaveeratitham P, Pensri P. Effect of flexibility exercise on lumbar angle: a study among non-specific low back pain patients. J Bodyw Mov Ther. 2012 Apr;16(2):236-43. doi: 10.1016/j.jbmt.2011.08.001. Epub 2011 Aug 31. PMID 22464123
- [Background] Lin N, Li Y, Bebawy JF, Dong J, Hua L. Abdominal circumference but not the degree of lumbar flexion affects the accuracy of lumbar interspace identification by Tuffier's line palpation method: an observational study. BMC Anesthesiol. 2015 Jan 21;15:9. doi: 10.1186/1471-2253-15-9. eCollection 2015. PMID 25670920
- [Background] Kopacz DJ, Neal JM, Pollock JE. The regional anesthesia "learning curve". What is the minimum number of epidural and spinal blocks to reach consistency? Reg Anesth. 1996 May-Jun;21(3):182-90. PMID 8744658
- [Background] Charuluxananan S, Kyokong O, Somboonviboon W, Pothimamaka S. Learning manual skills in spinal anesthesia and orotracheal intubation: is there any recommended number of cases for anesthesia residency training program? J Med Assoc Thai. 2001 Jun;84 Suppl 1:S251-5. PMID 11529340
- [Background] Smith MP, Sprung J, Zura A, Mascha E, Tetzlaff JE. A survey of exposure to regional anesthesia techniques in American anesthesia residency training programs. Reg Anesth Pain Med. 1999 Jan-Feb;24(1):11-6. doi: 10.1016/s1098-7339(99)90159-1. PMID 9952089
- [Background] Whitty R, Moore M, Macarthur A. Identification of the lumbar interspinous spaces: palpation versus ultrasound. Anesth Analg. 2008 Feb;106(2):538-40, table of contents. doi: 10.1213/ane.0b013e31816069d9. PMID 18227313
- [Background] Tanaka K, Irikoma S, Kokubo S. Identification of the lumbar interspinous spaces by palpation and verified by X-rays. Braz J Anesthesiol. 2013 May-Jun;63(3):245-8. doi: 10.1016/S0034-7094(13)70224-1. English, Portuguese, Spanish. PMID 23683445
- [Background] Mosaffa F, Karimi K, Madadi F, Khoshnevis SH, Daftari Besheli L, Eajazi A. Post-dural Puncture Headache: A Comparison Between Median and Paramedian Approaches in Orthopedic Patients. Anesth Pain Med. 2011 Fall;1(2):66-9. doi: 10.5812/kowsar.22287523.2159. Epub 2011 Sep 26. PMID 25729658
- [Background] Amorim JA, Gomes de Barros MV, Valenca MM. Post-dural (post-lumbar) puncture headache: risk factors and clinical features. Cephalalgia. 2012 Sep;32(12):916-23. doi: 10.1177/0333102412453951. Epub 2012 Jul 27. PMID 22843225
- [Background] Srivastava V, Jindal P, Sharma JP. Study of post dural puncture headache with 27G Quincke & Whitacre needles in obstetrics/non obstetrics patients. Middle East J Anaesthesiol. 2010 Jun;20(5):709-17. PMID 20803861
- [Background] Chan ST. Incidence of back pain after lumbar epidural anaesthesia for non-obstetric surgery--a preliminary report. Med J Malaysia. 1995 Sep;50(3):241-5. PMID 8926902
- [Background] Snijders CJ, Hermans PF, Kleinrensink GJ. Functional aspects of cross-legged sitting with special attention to piriformis muscles and sacroiliac joints. Clin Biomech (Bristol). 2006 Feb;21(2):116-21. doi: 10.1016/j.clinbiomech.2005.09.002. Epub 2005 Nov 2. PMID 16260074